CLINICAL TRIAL: NCT04357275
Title: The RIsk Stratification in COVID-19 Patients in the ICU Registry
Acronym: RISC-19-ICU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-req-2020-00322
Record Dates: First submitted 2020-04-15; First posted 2020-04-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Critical Illness; ARDS; Inflammatory Response; COVID-19; Circulatory Shock
MeSH Terms: conditions — Critical Illness; COVID-19; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU admissions due to COVID-19
  Interventions: Other: ICU treatment

INTERVENTIONS:
Other: ICU treatment — ICU treatment according to standard of care

SUMMARY:
The Risk stratification in COVID-19 patients in the ICU (RISC-19-ICU) registry was founded during the emerging SARS-CoV-2 pandemic. COVID-19 is a novel disease caused by infection with the SARS-CoV-2 virus that was first described in December 2019. The disease has spread exponentially in many countries and has reached global pandemic status within three months. According to first experience, hospitalization was required in approximately 20 % of cases and severe, life-threatening illness resulted in approximately 10 %. In some countries, health care systems were overwhelmed by the rapid increase in critically ill patients that far exceeded their capacity. It is thus of utmost importance to gain knowledge about the characteristics and course of critically ill patients with COVID-19 and to stratify these patients according to their risk for further deterioration. A key part of fighting this pandemic is to exchange scientific information and advance our understanding of the disease.

The Risk stratification in COVID-19 patients in the ICU (RISC-19-ICU) registry aims to collect an anonymized dataset to characterize patients that develop life-threatening critical illness due to COVID-19 and make it accessible to collaborative analysis.

The data collected may be composed of a core dataset and/or an extended dataset. The core dataset consists of a basic set of parameters, of which many are commonly generated during treatment of critically ill patients with COVID-19 in an intensive care unit (the individual parameters are marked yellow in the attached case report forms, and are clearly marked on the electronic case report forms during data entry). The extended dataset consists of parameters that may be measured during treatment of critically ill patients with COVID-19 in an intensive care unit, depending on clinical practice, indication and availability of the measurement method. The data accumulating in the registry as the pandemic or subsequent waves develop are made available to the collaborators to support an optimal response to the pandemic threat. The information gained on the initial characteristics and disease course via the RISC-19-ICU registry may contribute to a better understanding of the risk factors for developing critical illness due to COVID-19 and for an unfavorable disease course, and thus support informed patient triage and management decisions.

Initial research questions are (I) to perform risk stratification of critically ill patients with COVID-19 to find predictors associated with the development of critical illness due to COVID-19: characterization of the study population, which are critically ill patients with COVID-19: inflammation, oxygenation, circulatory function, among other parameters collected in the registry, and (II) to perform risk stratification of critically ill patients with COVID-19 to predict outcome after ICU admission (ICU mortality, ICU length of stay): characterization of patients grouped by disease course in the ICU, based on inflammation, oxygenation, circulatory function, and other parameters collected in the registry.

ELIGIBILITY:
Inclusion Criteria:

* Admission to an intensive care unit in a collaborating center due to COVID-19

Exclusion Criteria:

* Missing ethical approval

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to an intensive care unit in a collaborating center due to COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | During inclusion period

SECONDARY OUTCOMES:
Hospital mortality | During inclusion period
ICU length of stay | During inclusion period

CONTACTS AND LOCATIONS:
Overall Officials: Matthias P Hilty, MD, Principal Investigator — RISC-19-ICU board; Pedro D Wendel Garcia, MSc, Study Chair — RISC-19-ICU board; Reto A Schüpbach, MD, Study Chair — RISC-19-ICU board; Jonathan Montomoli, MD, PhD, Study Chair — RISC-19-ICU board; Philippe Guerci, MD, Study Chair — RISC-19-ICU board; Theirry Fumeaux, MD, Study Chair — RISC-19-ICU board
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
* Each collaborator's data is available for their own use
  * The collaborators are encouraged to share their analysis code (the standard is R code)
  * Analysis on the entire registry dataset may be performed using the same analysis pathway. To request analysis on the entire dataset, a protocol may be submitted to the board
  * The board may make some descriptive data publicly available to support the coordination of the response to the pandemic threat
  * Scientific findings will be jointly published in a scientific journal according to a collaboration agreement

REFERENCES:
- [Derived] Wendel-Garcia PD, Moser A, Jeitziner MM, Aguirre-Bermeo H, Arias-Sanchez P, Apolo J, Roche-Campo F, Franch-Llasat D, Kleger GR, Schrag C, Pietsch U, Filipovic M, David S, Stahl K, Bouaoud S, Ouyahia A, Fodor P, Locher P, Siegemund M, Zellweger N, Cereghetti S, Schott P, Gangitano G, Wu MA, Alfaro-Farias M, Vizmanos-Lamotte G, Ksouri H, Gehring N, Rezoagli E, Turrini F, Lozano-Gomez H, Carsetti A, Rodriguez-Garcia R, Yuen B, Weber AB, Castro P, Escos-Orta JO, Dullenkopf A, Martin-Delgado MC, Aslanidis T, Perez MH, Hillgaertner F, Ceruti S, Franchitti Laurent M, Marrel J, Colombo R, Laube M, Fogagnolo A, Studhalter M, Wengenmayer T, Gamberini E, Buerkle C, Buehler PK, Keiser S, Elhadi M, Montomoli J, Guerci P, Fumeaux T, Schuepbach RA, Jakob SM, Que YA, Hilty MP; RISC-19-ICU Investigators. Dynamics of disease characteristics and clinical management of critically ill COVID-19 patients over the time course of the pandemic: an analysis of the prospective, international, multicentre RISC-19-ICU registry. Crit Care. 2022 Jul 4;26(1):199. doi: 10.1186/s13054-022-04065-2. PMID 35787726
- [Derived] Hilty MP, Moser A, David S, Wendel Garcia PD, Capaldo G, Keiser S, Fumeaux T, Guerci P, Montomoli J, Van Boeckel TP, Jeitziner MM, Que YA, Jakob S, Schupbach RA; RISC-19-ICU Investigators for Switzerland. Near real-time observation reveals increased prevalence of young patients in the ICU during the emerging third SARS-CoV-2 wave in Switzerland. Swiss Med Wkly. 2021 Jul 21;151:Swiss Med Wkly. 2021;151:w20553. doi: 10.4414/smw.2021.20553. eCollection 2021 Jul 19. PMID 34291810